CLINICAL TRIAL: NCT05127135
Title: A Study to Evaluate the Safety and Clinical Activity of Allogeneic CAR-T Targeting CD7 in Patients With Refractory or Relapsed T Cell Malignancies
Brief Title: Safety and Efficacy of ThisCART7 in Patients With Refractory or Relapsed T Cell Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundamenta Therapeutics, Ltd. (Industry)
Collaborators: The First Affiliated Hospital of University of Science and Technology of China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ThisCART7
Record Dates: First submitted 2021-11-09; First posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: T-Acute Lymphoblastic Leukemia; T-cell Non-Hodgkin Lymphoma; T-cell Acute Lymphoblastic Lymphoma
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ThisCART7 cells injections (Experimental): In this study, allogeneic anti-CD7 CAR T Cells(ThisCART7 cells) is used to treat patients with refractory or relapsed CD7 positive T cell malignancies.
  Interventions: Biological: ThisCART7 cells

INTERVENTIONS:
Biological: ThisCART7 cells — 0.5-6 x 10^6 CAR T cells per kg body weight

SUMMARY:
This is a single dose escalation study to evaluate the safety and clinical activity of ThisCART7(Allogeneic CAR-T targeting CD7) in patients with refractory or relapsed CD7 positive T cell malignancies.

DETAILED DESCRIPTION:
This is a single-center, nonrandomized, open-label, dose-escalation study to evaluate the safety and clinical activity of ThisCART7 in patients with refractory or relapsed CD7 positive T cell malignancies, such as T-cell Acute Lymphoblastic Leukemia, T-cell Acute Lymphoblastic Lymphoma and T-cell Non-Hodgkin Lymphoma. The dose range is 0.5-6 x 10^6 cells per kg body weight.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with relapsed and refractory CD7 + T cell hematologic malignancies (including, but not limited to, T-cell leukemia, extranodal NK/ T-cell lymphoma nasal, peripheral T-cell lymphoma, enteropathy associated T-cell lymphoma and anaplastic T-cell lymphoma, etc.);
2. No alternative treatment options deemed by investigator;
3. Measurable or detectble disease at time of enrollment;
4. Age 18-70 years old, no gender and race limited;
5. Eastern cooperative oncology group (ECOG) performance status of ≤2;
6. Cardiac ejection fraction ≥ 40%, no evidence of pericardial effusion as determined by an echocardiogram (ECHO);
7. Estimated life expectancy > 12 weeks deemed by investigator;
8. Serum creatinine ≤ 1.5 upper limit of normal (ULN);
9. Serum ALT/ AST ≤ 5 upper limit of normal (ULN);
10. Signed informed consent form (ICF).

Exclusion Criteria:

1. Women in pregnancy or lactation;
2. Uncontrolled infection;
3. Active hepatitis B virus or hepatitis C virus infection;
4. Concurrent use of corticosteroids or other immunosuppressant medications for chronic disease;
5. Prior treatment with an allogeneic stem cell transplant within 100 days;
6. Grade 2-4 Active graft versus host disease;
7. History of HIV infection;
8. With central nervous system involvement;
9. Patients combine with other disease cause neutrophil count (ANC) < 750/uL or PLT< 50,000/uL.

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-01-22 (Actual); Primary Completion 2023-01-24 (Estimated); Study Completion 2023-12-24 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-related grade≥3Adverse Events or SAE | within 4 weeks after infusion
  Therapy-related adverse events or SAE will be recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0).

SECONDARY OUTCOMES:
Objective Response Rate | 4 to 6 weeks after infusion
  Description:
  For T-ALL, Objective response rate(ORR) is the percentage of patients who achieve CR or CRi, determined by National Comprehensive Cancer Network (NCCN) clinical practice guidelines in oncology Acute Lymphoblastic Leukemia (2020.V1) ;
  For lymphoma, ORR is the incidence of either a complete response (CR) or a partial response (PR). Response will be assessed using the 2014 Lugano criteria.

OTHER OUTCOMES:
Progression free survival time | 3 years
  The interval between administration and disease progression or death.
Overall survival time | 3 years
  The interval between administration and death caused by any reason.
Event-free survival | 3 years
  EFS is calculated from administration to death, progression of the disease, relapse or gene recurrence, whichever comes first, or last visit.

CONTACTS AND LOCATIONS:
Overall Officials: Wang Xingbing, Principal Investigator — The First Affiliated Hospital of USTC (Anhui Provincial Hospital)
Locations (2):
- China (2):
  - The First Affiliated Hospital of USTC (Anhui Provincial Hospital), Hefei, Anhui
  - Fundamenta Therapeutice Co.,Ltd, Suzhou, Jiangsu

IPD SHARING:
Plan to Share IPD: No